CLINICAL TRIAL: NCT02371369
Title: A Double-blind, Randomized, Placebo-controlled Phase 3 Study of Orally Administered PLX3397 in Subjects With Pigmented Villonodular Synovitis or Giant Cell Tumor of the Tendon Sheath
Brief Title: Phase 3 Study of Pexidartinib for Pigmented Villonodular Synovitis (PVNS) or Giant Cell Tumor of the Tendon Sheath (GCT-TS)
Acronym: ENLIVEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PLX108-10; 2014-000148-14 (EudraCT Number)
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Results first posted 2020-01-10 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-04

CONDITIONS: Pigmented Villonodular Synovitis; Giant Cell Tumors of the Tendon Sheath; Tenosynovial Giant Cell Tumor
Keywords: PLX3397; Pexidartinib; Colony Stimulating Factor 1 Receptor (CSF-1R) inhibitor
MeSH Terms: conditions — Synovitis, Pigmented Villonodular; Giant Cell Tumor of Tendon Sheath | interventions — pexidartinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) in Part 1, Open-label (no masking) in Part 2
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Part 1 - Pexidartinib (Experimental): Participants received blinded treatment of pexidartinib,1000 mg (5 capsules per day ) for 2 weeks, then 800 mg (4 capsules per day) for 22 weeks
  Interventions: Drug: Pexidartinib
- Part 1 - Placebo (Placebo Comparator): Participants received blinded treatment of matching placebo (5 capsules per day) for 2 weeks, then matching placebo (4 capsules per day) for 22 weeks
  Interventions: Drug: Placebo
- Part 2 - All Pexidartinib (Experimental): Participants received pexidartinib in Part 1 and in Part 2 at their prescribed dose
  Interventions: Drug: Pexidartinib
- Part 2 - Placebo-Pexidartinib (Experimental): Participants received placebo in Part 1 and pexidartinib in Part 2 at their prescribed dose
  Interventions: Drug: Pexidartinib; Drug: Placebo

INTERVENTIONS:
Drug: Pexidartinib — Each capsule contains 200 mg of pexidartinib for oral administration
  Other Names: PLX3397; Pexidartinib hydrochloride (HCl)
  Arms: Part 1 - Pexidartinib; Part 2 - All Pexidartinib; Part 2 - Placebo-Pexidartinib
Drug: Placebo — Placebo capsule matching pexidartinib capsule for oral administration
  Other Names: Placebo Capsule
  Arms: Part 1 - Placebo; Part 2 - Placebo-Pexidartinib

SUMMARY:
This is a Phase 3 clinical study, which aims to evaluate the effectiveness of an investigational drug called pexidartinib for the treatment of certain tumors for which surgical removal could cause more harm than good.

The main purpose of this study is to gather information about the investigational drug pexidartinib, which may help to treat tumors of pigmented villonodular synovitis (PVNS) or giant cell tumor of the tendon sheath (GCT-TS).

The study consists of two parts with a follow-up period. In Part 1, eligible study participants will be assigned to receive either pexidartinib or matching placebo for 24 weeks. A number of assessments will be carried out during the course of the study, including physical examinations, blood tests, imaging studies, electrocardiograms, and questionnaires. MRI scans will be used to evaluate the response of the tumors to the treatment. Some subjects, assigned to placebo in Part 1 transitioned to pexidartinib for Part 2.

Then a protocol amendment was written to allow only pexidartinib patients to continue into Part 2. Part 2 is a long-term treatment phase in which all participants receive open-label pexidartinib. There was also a follow-up period added to Part 2.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years.
2. A diagnosis of PVNS or GCT-TS (i) that has been histologically confirmed either by a pathologist at the treating institution or a central pathologist, and (ii) where surgical resection would be associated with potentially worsening functional limitation or severe morbidity (locally advanced disease), with morbidity determined consensually by qualified personnel (eg, two surgeons or a multi-disciplinary tumor board).
3. Measurable disease of at least 2 cm and otherwise based on RECIST 1.1, assessed from MRI scans by a central radiologist.
4. Symptomatic disease because of active PVNS or GCT-TS, defined as one or more of the following:

   1. a worst pain of at least 4 at any time during the week preceding the Screening Visit (based on scale of 0 to 10, with 10 representing "pain as bad as you can imagine").
   2. a worst stiffness of at least 4 at any time during the week preceding the Screening Visit (based on a scale of 0 to 10, with 10 representing "stiffness as bad as you can imagine").
5. Stable prescription of analgesic regimen during the 2 weeks prior to randomization.
6. During the 2 weeks prior to randomization, at least 4 of 7 consecutive days of Brief Pain Inventory (BPI) Worst Pain Numeric Rating Scale (NRS) items and Worst Stiffness NRS items completed correctly.
7. Women of childbearing potential must have a negative serum pregnancy test within the 14-day period prior to randomization. (Where demanded by local regulations, this test may be required within 72 hours of randomization.)
8. Males and females of childbearing potential are permitted in the study so long as they consent to avoid getting their partner pregnant or becoming pregnant, respectively, by using a highly effective contraception method, as described below, throughout the study and for up to 90 days after completion. Highly effective methods of contraception include: intra-uterine device (non-hormonal or hormonal), bilateral tubal occlusion, vasectomy, sexual abstinence, or barrier methods (eg, condom, diaphragm) used in combination with hormonal methods associated with inhibition of ovulation. Women of non-childbearing potential may be included if they are either surgically sterile or have been postmenopausal for ≥ 1 year. Women who have documentation of at least 12 months of spontaneous amenorrhea and have a follicle stimulating hormone (FSH) level > 40 milli-International units (mIU/mL) will be considered postmenopausal.
9. Adequate hematologic, hepatic, and renal function, defined by:

   * Absolute neutrophil count ≥ 1.5 × 10^9/L
   * aspartate aminotransferase/alanine (AST/ALT) ≤ 1.5 × upper limit of normal (ULN)
   * Hemoglobin > 10 g/dL
   * Total bilirubin ≤ 1.5 × ULN
   * Platelet count ≥ 100 × 10^9/L
   * Serum creatinine ≤ 1.5 × ULN
10. Willingness and ability to complete the Worst Pain NRS item, Worst Stiffness NRS item, Patient-reported Outcomes Measurement Information System (PROMIS) Physical Function Scale, and other self-assessment instruments throughout the study.
11. Willingness and ability to use an electronic diary.
12. Willingness and ability to provide written informed consent prior to any study-related procedures and to comply with all study requirements.

Exclusion Criteria

1. Investigational drug use within 28 days of randomization.
2. Previous use of pexidartinib or any biologic treatment targeting CSF-1 or the CSF-1R; previous use of oral tyrosine kinase inhibitors, eg, imatinib or nilotinib, are allowed.
3. Active cancer (either concurrent or within the last year of starting study treatment) that requires therapy (eg, surgical, chemotherapy, or radiation therapy), with the exception of adequately treated basal or squamous cell carcinoma of the skin, melanoma in-situ, carcinoma in-situ of the cervix or breast, or prostate carcinoma with a prostate-specific antigen value <0.2 ng/mL.
4. Known metastatic PVNS/GCT-TS.
5. Active or chronic infection with hepatitis C virus (HCV) or hepatitis B virus or known active or chronic infection with human immunodeficiency virus.
6. Known active tuberculosis.
7. Significant concomitant arthropathy in the affected joint, serious illness, uncontrolled infection, or a medical or psychiatric history that, in the Investigator's opinion, would likely interfere with the person's study participation or the interpretation of his or her results.
8. Women who are breastfeeding.
9. A screening Fridericia corrected QT interval (QTcF) ≥ 450 ms (men) or ≥ 470 ms (women).
10. MRI contraindications.
11. History of hypersensitivity to any excipients in the investigational product.
12. Inability to swallow capsules.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Team Leader, Study Director — Daiichi Sankyo
Locations (39):
- United States (19):
  - Mayo Clinic, Scottsdale, Arizona
  - University of Southern California, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - UCLA Medical Center, Santa Monica, California
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - : Dana Farber Cancer Institute, Boston, Massachusetts
  - Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - MD Anderson Cancer Center at Cooper, Camden, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke Cancer Center, Durham, North Carolina
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (3):
  - Chris O'Brien Lifehouse, Sydney, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Herlev Hospital, Herlev, Denmark
- France (2):
  - Centre Leon Bérard, Lyon
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Universitätsklinikum Essen, Essen
- Military Hospital-State Health Center, Budapest, Hungary
- Italy (2):
  - Istituto Ortopedico Rizzoli, Bologna, BO
  - Istituto Nazionale Tumori-Fondazione IRCCS, Milan, MI
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Radboud Univ. Medical Center, Nijmegen
- Centrum Onkologii-Instytut im. Marii Skłodowskiej-Curie, Warsaw, Poland
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Virgen del Rocío, Seville
- United Kingdom (2):
  - University College Hospital, London
  - The Royal Marsden NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Healey JH, Tap WD, Gelhorn HL, Ye X, Speck RM, Palmerini E, Stacchiotti S, Desai J, Wagner AJ, Alcindor T, Ganjoo K, Martin-Broto J, Wang Q, Shuster D, Gelderblom H, van de Sande M. Pexidartinib Provides Modest Pain Relief in Patients With Tenosynovial Giant Cell Tumor: Results From ENLIVEN. Clin Orthop Relat Res. 2023 Jan 1;481(1):107-116. doi: 10.1097/CORR.0000000000002335. Epub 2022 Aug 24. PMID 36001000
- [Derived] Lewis JH, Gelderblom H, van de Sande M, Stacchiotti S, Healey JH, Tap WD, Wagner AJ, Pousa AL, Druta M, Lin CC, Baba HA, Choi Y, Wang Q, Shuster DE, Bauer S. Pexidartinib Long-Term Hepatic Safety Profile in Patients with Tenosynovial Giant Cell Tumors. Oncologist. 2021 May;26(5):e863-e873. doi: 10.1002/onco.13629. Epub 2020 Dec 24. PMID 33289960
- [Derived] Tap W. ENLIVEN study: Pexidartinib for tenosynovial giant cell tumor (TGCT). Future Oncol. 2020 Sep;16(25):1875-1878. doi: 10.2217/fon-2020-0307. Epub 2020 Aug 5. PMID 32755241
- [Derived] Tap WD, Gelderblom H, Palmerini E, Desai J, Bauer S, Blay JY, Alcindor T, Ganjoo K, Martin-Broto J, Ryan CW, Thomas DM, Peterfy C, Healey JH, van de Sande M, Gelhorn HL, Shuster DE, Wang Q, Yver A, Hsu HH, Lin PS, Tong-Starksen S, Stacchiotti S, Wagner AJ; ENLIVEN investigators. Pexidartinib versus placebo for advanced tenosynovial giant cell tumour (ENLIVEN): a randomised phase 3 trial. Lancet. 2019 Aug 10;394(10197):478-487. doi: 10.1016/S0140-6736(19)30764-0. Epub 2019 Jun 19. PMID 31229240
- [Derived] Gelhorn HL, Tong S, McQuarrie K, Vernon C, Hanlon J, Maclaine G, Lenderking W, Ye X, Speck RM, Lackman RD, Bukata SV, Healey JH, Keedy VL, Anthony SP, Wagner AJ, Von Hoff DD, Singh AS, Becerra CR, Hsu HH, Lin PS, Tap WD. Patient-reported Symptoms of Tenosynovial Giant Cell Tumors. Clin Ther. 2016 Apr;38(4):778-93. doi: 10.1016/j.clinthera.2016.03.008. Epub 2016 Apr 1. PMID 27041409

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part 1 was a double-blind, randomized, Pexidartinib or placebo in participants with symptomatic TGCT for whom surgical resection would be associated with potentially worsening functional limitation or severe morbidity. Part 2 is a long-term treatment phase in which all eligible participants received open-label Pexidartinib.
Pre-assignment Details: Participants were screened for inclusion and exclusion criteria. Screening procedures were performed after consent was obtained and within the 42 days before the first dose of study drug, unless otherwise noted.
Groups:
- Pexidartinib Part 1, Then Pexidartinib Part 2: Participants received Pexidartinib,1000 mg (5 capsules per day ) for 2 weeks, then 800 mg (4 capsules per day) for 22 weeks in Part 1 of study. Eligible participants from this group also received Pexidartinib in Part 2 at their prescribed dose.
  Pexidartinib: Each capsule contains 200 mg of pexidartinib for oral administration.
- Placebo Part 1, Then Pexidartinib Part 2: Participants received treatment of matching placebo (5 capsules per day) for 2 weeks, then matching placebo (4 capsules per day) for 22 weeks in Part 1 of study. Eligible participants from this group also received Pexidartinib in Part 2 at their prescribed dose.
  Placebo: Placebo capsule matching Pexidartinib capsule for oral administration. Pexidartinib: Each capsule contains 200 mg of Pexidartinib for oral administration (Part 2).
Period: Part 1
Arm/Group | Pexidartinib Part 1, Then Pexidartinib Part 2 | Placebo Part 1, Then Pexidartinib Part 2
Started | 61 | 59
Completed | 52 | 48
Not Completed | 9 | 11
Not completed — Physician Decision | 0 | 3
Not completed — Adverse Event | 8 | 0
Not completed — Withdrawal by Subject | 1 | 6
Not completed — Disease progression | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Part 2
Arm/Group | Pexidartinib Part 1, Then Pexidartinib Part 2 | Placebo Part 1, Then Pexidartinib Part 2
Started | 48 (N=48; Only participants who were eligible to receive treatment in Part 2.) | 30 (N=30; Only participants who were eligible to receive treatment in Part 2.)
Completed | 0 | 0
Not Completed | 48 | 30
Not completed — Adverse Event | 6 | 5
Not completed — Withdrawal by Subject | 16 | 6
Not completed — Investigator decision | 1 | 2
Not completed — Death | 0 | 1
Not completed — Disease progression | 1 | 0
Not completed — Subject Noncompliance | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Subject transitioned to commercial supply | 6 | 4
Not completed — Subject transitioned to another DS pexidartinib protocol | 15 | 9
Not completed — Surgical resection of tumor | 1 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pexidartinib Part 1, Then Pexidartinib Part 2 | Placebo Part 1, Then Pexidartinib Part 2 | Total
Number analyzed (Participants) | 61 | 59 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 56 | 113
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (13.2) | 44.3 (13.6) | 44.5 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 71
  Male | 26 | 23 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 3 | 1 | 4
  White | 52 | 54 | 106
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 3 | 5
  Netherlands | 7 | 4 | 11
  Hungary | 2 | 1 | 3
  United States | 23 | 22 | 45
  Denmark | 1 | 2 | 3
  Poland | 2 | 0 | 2
  Italy | 8 | 9 | 17
  United Kingdom | 0 | 1 | 1
  Australia | 5 | 7 | 12
  France | 2 | 5 | 7
  Germany | 4 | 2 | 6
  Spain | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Symptomatic, Locally Advanced Tenosynovial Giant Cell Tumor (TGCT) Achieving Complete or Partial Response to Pexidartinib Compared With That of Placebo Per Response Evaluation Criteria in Solid Tumors Version 1.1 at Week 25
Description: Complete response (CR) and partial responses (PR) were assessed based on centrally-read magnetic resonance imaging (MRI) scans and Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1). A CR was defined as disappearance of all tumors and a PR was defined as at least a 30% decrease in the sum of diameters of target tumors using the baseline sum diameters as the reference.
Time Frame: Week 25
Population: Best overall response was assessed in the Intent-to-Treat (ITT) population.
Measure: Number; unit: Percentage of participants
Groups:
- Pexidartinib Part 1: Participants received treatment of Pexidartinib,1000 mg (5 capsules per day ) for 2 weeks, then 800 mg (4 capsules per day) for 22 weeks Pexidartinib: Each capsule contains 200 mg of Pexidartinib for oral administration.
- Placebo Part 1: Participants received treatment of matching placebo (5 capsules per day) for 2 weeks, then matching placebo (4 capsules per day) for 22 weeks Placebo: Placebo capsule matching Pexidartinib capsule for oral administration.
Arm/Group | Pexidartinib Part 1 | Placebo Part 1
Number analyzed (Participants) | 61 | 59
Percentage of participants
  Complete Response (CR) | 14.8 | 0
  Partial Response (PR) | 24.6 | 0
  Response (CR or PR) | 39.3 | 0
Statistical Analysis 1: Comparison: Pexidartinib Part 1 vs Placebo Part 1; Treatment comparison between the pexidartinib and placebo groups at Week 25; Test type: Other — Treatment comparison analysis; p < 0.0001, Fisher's Exact Test

2. Secondary Outcome: Mean Change From Baseline For Range of Motion (ROM) Score in Participants Receiving Pexidartinib Compared With Those on Placebo Up to Week 25
Description: Range of motion (ROM) of the joint was assessed by a qualified, independent, and blinded or third-party assessors at the clinical site. Measurements were recorded in degrees. At baseline, the plane of movement with the smallest relative value (worst) was identified and this plane was used for evaluating the relative change of motion subsequently. Only the plane with the worst impaired ROM at baseline was selected for subsequent analyses.
Time Frame: Baseline, Week 13, and Week 25
Population: Range of motion was assessed in the ITT population in participants where data were available.
Measure: Least Squares Mean (Standard Error); unit: degrees
Arm/Group | Pexidartinib Part 1 | Placebo Part 1
Number analyzed (Participants) | 61 | 59
degrees
  Baseline: number analyzed (Participants) | 61 | 58
  Baseline | 62.5 (3.2) | 62.9 (2.9)
  Week 13: number analyzed (Participants) | 52 | 53
  Week 13 | 13.0 (2.3) | 4.8 (2.6)
  Week 25: number analyzed (Participants) | 45 | 43
  Week 25 | 15.1 (2.1) | 6.2 (2.4)
Statistical Analysis 1: Comparison: Pexidartinib Part 1 vs Placebo Part 1; Treatment comparison between the pexidartinib and placebo groups at Week 25; Test type: Other — Treatment comparison analysis; p = 0.0043, Fisher's Exact Test

3. Secondary Outcome: Percentage of Participants With Symptomatic, Locally Advanced Tenosynovial Giant Cell Tumor (TGCT) Achieving Complete or Partial Response Based on Tumor Volume Score (TVS) After Receiving Pexidartinib Compared With Those on Placebo at Week 25
Description: Complete response (CR) and partial response (PR) were assessed using tumor volume score (TVS). A CR was defined as disappearance of all tumors and a PR was defined as at least a 30% decrease in the sum of diameters of target tumors using the baseline sum diameters as the reference. TVS is a semi-quantitative MRI scoring system that describes tumor mass and is based on 10% increments of the estimated volume of the maximally distended synovial cavity or tendon sheath involved. A tumor that is equal in volume to that of a maximally distended synovial cavity or tendon sheath was scored 10; a score of 0 indicated no evidence of tumor.
Time Frame: Week 25
Population: Best overall response was assessed in the ITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Pexidartinib Part 1 | Placebo Part 1
Number analyzed (Participants) | 61 | 59
Percentage of participants
  Complete Response (CR) | 4.9 | 0
  Partial Response (PR) | 50.8 | 0
  Response (CR or PR) | 55.7 | 0
Statistical Analysis 1: Comparison: Pexidartinib Part 1 vs Placebo Part 1; Treatment comparison between the pexidartinib and placebo groups at Week 25; Test type: Other — Treatment comparison analysis; p < 0.0001, Fisher's Exact Test

4. Secondary Outcome: Mean Change From Baseline in the Patient-reported Outcomes Measurement Information System (PROMIS) Physical Function Score in Participants Receiving Pexidartinib Compared With Those on Placebo Up to Week 25
Description: The Patient-reported Outcomes Measurement Information System (PROMIS) physical function scale was used to assess physical function of the upper and lower limbs. The scale ranged from 1 defined as 'unable to do' or 'cannot do' to 5 defined as 'without any difficulty' or 'not at all', where higher scores represent better outcomes.
Time Frame: at Week 9 , Week 17, and Week 25
Population: Physical function was assessed in the ITT population in participants where data were available.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pexidartinib Part 1 | Placebo Part 1
Number analyzed (Participants) | 61 | 59
units on a scale
  Week 9: number analyzed (Participants) | 38 | 41
  Week 9 | 2.8 (1.0) | -0.4 (0.8)
  Week 17: number analyzed (Participants) | 39 | 40
  Week 17 | 3.2 (1.1) | 0.2 (1.0)
  Week 25: number analyzed (Participants) | 38 | 31
  Week 25 | 4.1 (1.1) | -0.9 (1.0)
Statistical Analysis 1: Comparison: Pexidartinib Part 1 vs Placebo Part 1; Treatment comparison between pexidartinib and placebo groups at Week 25; Test type: Other — Treatment comparison analysis; p = 0.0019, Mixed effects model for repeated measure

5. Secondary Outcome: Mean Change From Baseline for Worst Stiffness Numeric Rating Scale Score (NRS) in Participants Receiving Pexidartinib Compared With Those on Placebo Up to Week 25
Description: The Worst Stiffness Numeric Rating Scale (NRS) was a 1-item, self-administered questionnaire assessing the "worst" stiffness in the last 24 hours. The NRS for this item ranged from 0 (no stiffness) to 10 (stiffness as bad as you can imagine).
Time Frame: Baseline, Week 9, Week 17, and Week 25
Population: Worst stiffness was assessed in the ITT population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Pexidartinib Part 1 | Placebo Part 1
Number analyzed (Participants) | 61 | 59
units on a scale
  Baseline: number analyzed (Participants) | 59 | 58
  Baseline | 5.6 (0.2) | 5.9 (0.3)
  Week 9: number analyzed (Participants) | 30 | 38
  Week 9 | -1.5 (0.3) | -0.5 (0.3)
  Week 17: number analyzed (Participants) | 37 | 30
  Week 17 | -2.4 (0.3) | -0.4 (0.3)
  Week 25: number analyzed (Participants) | 33 | 35
  Week 25 | -2.5 (0.3) | -0.3 (0.3)
Statistical Analysis 1: Comparison: Pexidartinib Part 1 vs Placebo Part 1; Treatment comparison between the pexidartinib and placebo groups at Week 25; Test type: Other — Treatment comparison analysis; p < 0.0001, Mixed effects model for repeated measure

6. Secondary Outcome: Percentage of Participants Who Responded With a Decrease of at Least 30% in the Mean Brief Pain Inventory Worst Pain Numeric Rating Scale Score Among Participants Receiving Pexidartinib Compared With Those on Placebo at Week 25
Description: The Brief Pain Inventory (BPI) Worst Pain Numeric Rating Scale Score (NRS) was a 1-item, self-administered questionnaire assessing the "worst" pain in the last 24 hours. The NRS for this item ranged from 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: Week 25
Population: Worst pain was assessed in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Pexidartinib Part 1 | Placebo Part 1
Number analyzed (Participants) | 61 | 59
percentage of participants | 31.1 | 15.3

7. Secondary Outcome: Number of Responders to Pexidartinib With and Without Disease Progression
Description: Duration of response (DOR) based on RECIST 1.1 is defined as the date of the first recorded response to the first date of documented disease progression. The overall number of responses and the number of participants with and without disease progression was assessed.
Time Frame: By Week 96
Population: The overall number of responses and the number of participants with and without disease progression were assessed in the ITT population, specifically among the Pexidartinib Part 1, Pexidartinib Part 2; Pexidartinib Part 2 only, All Pexidartinib Treated participants, . Participants randomized to Placebo Part 1 only were not analyzed.
Measure: Number; unit: participants
Groups:
- Pexidartinib Part 1 and Part 2: Part 1: Participants received treatment of pexidartinib,1000 mg (5 capsules per day ) for 2 weeks, then 800 mg (4 capsules per day) for 22 weeks
  Part 2: Participants also received pexidartinib at their prescribed dose.
  Pexidartinib: Each capsule contains 200 mg of pexidartinib for oral administration
- Placebo Part 1, Pexidartinib Part 2: Participants that received placebo in part 1 and received Pexidartinib in Part 2 at their prescribed dose.
  Pexidartinib: Each capsule contains 200 mg of pexidartinib for oral administration
- All Pexidartinib Treated: All participants who received Pexidartinib in Part 1 and Part 2 as well as those who only received Pexidartinib in Part 2.
Arm/Group | Pexidartinib Part 1 and Part 2 | Placebo Part 1, Pexidartinib Part 2 | All Pexidartinib Treated
Number analyzed (Participants) | 61 | 30 | 91
participants
  Number of responses | 23 | 12 | 35
  Week 12 (Day 84); Without disease progression | 23 | 12 | 35
  Week 12 (Day 84); With disease progression | 0 | 0 | 0
  Week 24 (Day 168); Without disease progression | 23 | 12 | 35
  Week 24 (Day 168); With disease progression | 0 | 0 | 0
  Week 48 (Day 336); Without disease progression | 15 | 9 | 24
  Week 48 (Day 336); With disease progression | 1 | 0 | 1
  Week 72 (Day 504); Without disease progression | 9 | 3 | 12
  Week 72 (Day 504); With disease progression | 1 | 0 | 1
  Week 96 (Day 672); Without disease progression | 2 | 1 | 3
  Week 96 (Day 672); With disease progression | 1 | 0 | 1

8. Secondary Outcome: Number of Responders to Pexidartinib With and Without Disease Progression Based on Tumor Volume Score
Description: Tumor Volume Score (TVS) is a semi-quantitative MRI scoring system that describes tumor mass and is based on 10% increments of the estimated volume of the maximally distended synovial cavity or tendon sheath involved. A tumor that is equal in volume to that of a maximally distended synovial cavity or tendon sheath was scored 10; a score of 0 indicated no evidence of tumor. The overall number of responses and the number of participants with and without disease progression was assessed.
Time Frame: By Week 120
Population: The overall number of responses and the number of participants with and without disease progression was assessed in the ITT population, specifically among the Pexidartinib Part 1, Pexidartinib Part 2; Pexidartinib Part 2 only; and All Pexidartinib Treated participants. Participants who received Placebo Part 1 only were not analyzed.
Measure: Number; unit: participants
Groups:
- Pexidartinib in Part 1 and Part 2: Participants received treatment of Pexidartinib,1000 mg (5 capsules per day ) for 2 weeks, then 800 mg (4 capsules per day) for 22 weeks in Part 1 and also received Pexidartinib in Part 2 at their prescribed dose.
  Pexidartinib: Each capsule contains 200 mg of pexidartinib for oral administration
- Placebo Part 1, Pexidartinib Part 2: Participants received treatment of matching placebo (5 capsules per day) for 2 weeks, then matching placebo (4 capsules per day) for 22 weeks in Part 1 and also received Pexidartinib in Part 2 at their prescribed dose.
  Placebo: Placebo capsule matching Pexidartinib capsule for oral administration Pexidartinib: Each capsule contains 200 mg of Pexidartinib for oral administration.
- All Pexidartinib Treated: All participants who received pexidartinib in Part 1 and Part 2 as well as those who received pexidartinib in Part 2 only.
Arm/Group | Pexidartinib in Part 1 and Part 2 | Placebo Part 1, Pexidartinib Part 2 | All Pexidartinib Treated
Number analyzed (Participants) | 61 | 30 | 91
participants
  Number of responders | 34 | 18 | 52
  Week 12 (Day 84); Without disease progression | 33 | 18 | 51
  Week 12 (Day 84); With disease progression | 0 | 0 | 0
  Week 24 (Day 168); Without disease progression | 32 | 18 | 50
  Week 24 (Day 168); With disease progression | 0 | 0 | 0
  Week 48 (Day 336); Without disease progression | 22 | 13 | 35
  Week 48 (Day 336); With disease progression | 3 | 1 | 4
  Week 72 (Day 504); Without disease progression | 13 | 3 | 16
  Week 72 (Day 504); With disease progression | 3 | 1 | 4
  Week 96 (Day 672); Without disease progression | 3 | 1 | 4
  Week 96 (Day 672); With disease progression | 3 | 1 | 4
  Week 120 (Day 840); Without disease progression | 1 | 0 | 1
  Week 120 (Day 840); With disease progression | 3 | 1 | 4

9. Secondary Outcome: Duration of Response (DOR) Based on RECIST 1.1
Description: Duration of response (DOR) based on RECIST 1.1 is defined from the date of the first recorded evidence of response to the first date of documented disease progression.
Time Frame: Date of first documentation of objective response up to date of first documentation of progressive disease, assessed up to end of study (approximately 71 months)
Population: DOR was assessed in the ITT population, specifically among the Pexidartinib Part 1, Pexidartinib Part 2; Pexidartinib Part 2 only. Participants randomized to Placebo Part 1 only were not analyzed. DOR was based on numbers of responders only.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pexidartinib Part 1 and Part 2 | Placebo Part 1, Pexidartinib Part 2
Number analyzed (Participants) | 37 | 18
months | NA [31.01 to NA] — Median and upper limit 95% CI was not estimable due to insufficient number of events. | NA [39.0 to NA] — Median and upper limit 95% CI was not estimable due to insufficient number of events.

10. Secondary Outcome: Duration of Response (DOR) Based on Tumor Volume Score (TVS)
Description: Duration of response (DOR) based on TVS is defined from the date of the first recorded evidence of response to the first date of documented disease progression.
Time Frame: as for outcome 9
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pexidartinib Part 1 and Part 2 | Placebo Part 1, Pexidartinib Part 2
Number analyzed (Participants) | 41 | 21
months | 52.70 [38.60 to NA] — Upper limit 95% CI was not estimable due to insufficient number of events. | NA [NA to NA] — Median and 95% CIs was not estimable due to insufficient number of events.

11. Secondary Outcome: Percentage of Participants Reporting Frequent (≥10%) Treatment-Emergent Adverse Events by Preferred Term
Description: Treatment-emergent adverse events (TEAEs) were defined as adverse events that started or worsened after the first dose of treatment and within 28 days after the last dose. The National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0 was used to grade adverse events. Any Grade and Grade ≥3 (severe) TEAEs are reported. TEAEs were coded using MedDRA version 17.1.
Time Frame: After the first dose of treatment up to 28 days after the last dose
Population: All safety events were assessed in the Safety Analysis Set.
Measure: Number; unit: Percentage of participants
Groups:
- Pexidartinib Part 1 and Part 2: Participants received treatment of Pexidartinib,1000 mg (5 capsules per day) for 2 weeks, then 800 mg (4 capsules per day) for 22 weeks and also received Pexidartinib in Part 2 at their prescribed dose.
  Pexidartinib: Each capsule contains 200 mg of Pexidartinib for oral administration.
Arm/Group | Pexidartinib Part 1 | Placebo Part 1 | Pexidartinib Part 1 and Part 2 | Placebo Part 1, Pexidartinib Part 2 | All Pexidartinib Treated
Number analyzed (Participants) | 61 | 59 | 61 | 30 | 91
Percentage of participants
  Any Hair color changes | 67.2 | 3.4 | 73.8 | 83.3 | 76.9
  Grade ≥3 Hair color changes | 0 | 0 | 0 | 0 | 0
  Any Pruritis | 9.8 | 3.4 | 16.4 | 20.0 | 17.6
  Grade ≥3 Pruritis | 0 | 0 | 1.6 | 0 | 1.1
  Any Rash maculopapular | 9.8 | 1.7 | 14.8 | 10.0 | 13.2
  Grade ≥3 Rash maculopapular | 0 | 0 | 1.6 | 0 | 1.1
  Any Pruritis generalized | 8.2 | 0 | 8.2 | 10.0 | 8.8
  Grade ≥3 Pruritis generalized | 0 | 0 | 0 | 0 | 0
  Any Erythema | 1.6 | 0 | 3.3 | 20.0 | 8.8
  Grade ≥3 Erythema | 0 | 0 | 0 | 0 | 0
  Any Dry skin | 3.3 | 3.4 | 6.6 | 10.0 | 7.7
  Grade ≥3 Dry skin | 0 | 0 | 0 | 3.3 | 1.1
  Any Photosensitivity reaction | 0 | 0 | 1.6 | 10.0 | 4.4
  Grade ≥3 Photosensitivity reaction | 0 | 0 | 0 | 0 | 0
  Any Nausea | 37.7 | 40.7 | 44.3 | 20.0 | 36.3
  Grade ≥3 Nausea | 0 | 0 | 0 | 0 | 0
  Any Diarrhea | 19.7 | 25.4 | 26.2 | 30.0 | 27.5
  Grade ≥3 Diarrhea | 0 | 0 | 0 | 0 | 0
  Any Vomiting | 19.7 | 5.1 | 23.0 | 6.7 | 17.6
  Grade ≥3 Vomiting | 1.6 | 0 | 1.6 | 0 | 1.1
  Any Abdominal Pain | 16.4 | 10.2 | 21.3 | 6.7 | 16.5
  Grade ≥3 Abdominal Pain | 0 | 0 | 0 | 0 | 0
  Any Dry mouth | 9.8 | 3.4 | 13.1 | 13.3 | 13.2
  Grade ≥3 Dry mouth | 0 | 0 | 0 | 0 | 0
  Any Constipation | 11.5 | 5.1 | 14.8 | 10.0 | 13.2
  Grade ≥3 Constipation | 0 | 0 | 0 | 0 | 0
  Any Stomatitis | 6.6 | 1.7 | 8.2 | 10.0 | 8.8
  Grade ≥3 Stomatitis | 0 | 0 | 0 | 0 | 0
  Any Fatigue | 54.1 | 35.6 | 55.7 | 26.7 | 46.2
  Grade ≥3 Fatigue | 0 | 0 | 0 | 0 | 0
  Any Edema peripheral | 13.1 | 3.4 | 16.4 | 20.0 | 17.6
  Grade ≥3 Edema peripheral | 0 | 0 | 0 | 0 | 0
  Any Face edema | 13.1 | 1.7 | 14.8 | 20.0 | 16.5
  Grade ≥3 Face edema | 0 | 0 | 1.6 | 3.3 | 2.2
  Any Asthenia | 9.8 | 5.1 | 11.5 | 20.0 | 14.3
  Grade ≥3 Asthenia | 0 | 0 | 0 | 0 | 0
  Any Pyrexia | 6.6 | 1.7 | 8.2 | 13.3 | 9.9
  Grade ≥ Pyrexia | 0 | 0 | 0 | 0 | 0
  Any AST increased | 39.3 | 0 | 44.3 | 16.7 | 35.2
  Grade ≥3 AST increased | 9.8 | 0 | 9.8 | 6.7 | 8.8
  Any ALT increased | 27.9 | 1.7 | 31.1 | 23.3 | 28.6
  Grade ≥3 ALT increased | 9.8 | 0 | 9.8 | 10.0 | 9.9
  Any ALP increased | 14.8 | 0 | 14.8 | 3.3 | 11.0
  Grade ≥3 ALP increased | 6.6 | 0 | 6.6 | 3.3 | 5.5
  Any LDH increased | 11.5 | 0 | 11.5 | 10.0 | 11.0
  Grade ≥3 LDH increased | 1.6 | 0 | 1.6 | 0 | 1.1
  Any Weight increased | 3.3 | 0 | 4.9 | 10.0 | 6.6
  Grade ≥3 Weight increased | 0 | 0 | 0 | 0 | 0
  Any Dysgeusia | 24.6 | 1.7 | 27.9 | 23.3 | 26.4
  Grade ≥3 Dysgeusia | 0 | 0 | 0 | 0 | 0
  Any Headache | 19.7 | 18.6 | 23.0 | 20.0 | 22.0
  Grade ≥3 Headache | 0 | 0 | 1.6 | 0 | 1.1
  Any Dizziness | 9.8 | 15.3 | 13.1 | 13.3 | 13.2
  Grade ≥3 Dizziness | 1.6 | 0 | 1.6 | 0 | 1.1
  Any Paresthesia | 1.6 | 1.7 | 8.2 | 10.0 | 8.8
  Grade ≥3 Paresthesia | 0 | 0 | 0 | 0 | 0
  Any Memory impairment | 0 | 1.7 | 1.6 | 10.0 | 4.4
  Grade ≥3 Memory impairment | 0 | 0 | 0 | 0 | 0
  Any Arthralgia | 23.0 | 25.4 | 27.9 | 30.0 | 28.6
  Grade ≥3 Arthralgia | 3.3 | 1.7 | 3.3 | 0 | 2.2
  Any Pain in extremity | 6.6 | 6.8 | 9.8 | 13.3 | 11.0
  Grade ≥3 Pain in extremity | 0 | 1.7 | 0 | 0 | 0
  Any Periorbital edema | 18.0 | 1.7 | 24.6 | 13.3 | 20.0
  Grade ≥3 Periorbital edema | 1.6 | 0 | 1.6 | 0 | 1.1
  Any Eyelid edema | 3.3 | 0 | 4.9 | 10.0 | 6.6
  Grade ≥3 Eyelid edema | 0 | 0 | 0 | 0 | 0
  Any Decreased appetite | 16.4 | 10.2 | 18.0 | 10.0 | 15.4
  Grade ≥3 Decreased appetite | 0 | 0 | 0 | 0 | 0
  Any Hypertension | 14.8 | 10.2 | 19.7 | 30.0 | 13.1
  Grade ≥3 Hypertension | 4.9 | 0 | 4.9 | 6.7 | 5.5
  Any Upper respiratory tract infection | 1.6 | 0 | 11.5 | 3.3 | 8.8
  Grade ≥3 Upper respiratory tract infection | 0 | 0 | 0 | 0 | 0
  Any Cough | 4.9 | 5.1 | 6.6 | 10.0 | 7.7
  Grade ≥3 Cough | 0 | 0 | 0 | 0 | 0
  Any Dyspnea | 1.6 | 0 | 4.9 | 10.0 | 7.7
  Grade ≥3 Dyspnea | 0 | 0 | 0 | 0 | 0
  Any Insomnia | 4.9 | 3.4 | 4.9 | 10.0 | 6.6
  Grade ≥3 Insomnia | 0 | 0 | 0 | 0 | 0
  Any Rash | 14.8 | 5.1 | 27.9 | 23.3 | 26.4
  Grade ≥3 Rash | 1.6 | 0 | 1.6 | 0 | 1.1

12. Other Pre Specified Outcome: Percentage of Participants With Symptomatic, Locally Advanced Tenosynovial Giant Cell Tumor (TGCT) Achieving Complete or Partial Response to Pexidartinib Compared With That of Placebo Per Response Evaluation Criteria in Solid Tumors Version 1.1 by Week 49
Description: Complete (CR) and partial responses (PR) were assessed based on centrally-read magnetic resonance imaging (MRI) scans and Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1). A CR was defined as disappearance of all tumors and a PR was defined as at least a 30% decrease in the sum of diameters of target tumors using the baseline sum diameters as the reference.
Time Frame: By Week 49
Population: Best overall response was assessed in the ITT population.
Measure: Number; unit: Percentage of participants
Arm/Group | Pexidartinib Part 1 and Part 2 | Placebo Part 1, Pexidartinib Part 2 | All Pexidartinib Treated
Number analyzed (Participants) | 61 | 30 | 91
Percentage of participants
  Complete Response (CR) | 24.6 | 23.3 | 24.2
  Partial Response (PR) | 29.5 | 30.0 | 29.7
  Response (CR or PR) | 54.1 | 53.3 | 53.8

13. Other Pre Specified Outcome: Mean Change From Baseline For Range of Motion (ROM) Score in Participants Receiving Pexidartinib Compared With Those on Placebo by Week 49
Description: as for outcome 2
Time Frame: By Week 49
Population: Range of Motion (ROM) was assessed in the ITT population.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Pexidartinib Part 1 and Part 2 | Placebo Part 1, Pexidartinib Part 2 | All Pexidartinib Treated
Number analyzed (Participants) | 61 | 30 | 91
degrees
  Baseline | 62.5 (24.8) | 66.5 (22.9) | 63.8 (24.2)
  Week 25: number analyzed (Participants) | 45 | 24 | 69
  Week 25 | 15.6 (14.9) | 13.1 (12.9) | 14.8 (14.2)
  Week 49: number analyzed (Participants) | 33 | 22 | 55
  Week 49 | 14.4 (19.5) | 12.0 (13.4) | 13.4 (17.3)

14. Other Pre Specified Outcome: Mean Change From Baseline in the Patient-reported Outcomes Measurement Information System (PROMIS) Physical Function Score in Participants Receiving Pexidartinib Compared With Those on Placebo by Week 49
Description: as for outcome 4
Time Frame: By Week 49
Population: Physical function was assessed in the ITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pexidartinib Part 1 and Part 2 | Placebo Part 1, Pexidartinib Part 2 | All Pexidartinib Treated
Number analyzed (Participants) | 61 | 30 | 91
units on a scale
  Week 25: number analyzed (Participants) | 38 | 16 | 54
  Week 25 | 3.6 (4.9) | 4.9 (6.3) | 4.0 (5.4)
  Week 49: number analyzed (Participants) | 25 | 14 | 39
  Week 49 | 4.7 (4.4) | 7.6 (6.3) | 5.8 (5.2)

15. Other Pre Specified Outcome: Mean Change From Baseline for Worst Stiffness Numeric Rating Scale Score (NRS) in Participants Receiving Pexidartinib Compared With Those on Placebo by Week 49
Description: as for outcome 5
Time Frame: Baseline, Week 25, and Week 49
Population: Worst stiffness was assessed in the ITT population, specifically among the Pexidartinib Part 1, Pexidartinib Part 2; Placebo Part 1, Pexidartinib Part 2; and All Pexidartinib Treated participants. Participants who received Placebo Part 1 only or Pexidartinib Part 2 only were not analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pexidartinib Part 1 and Part 2 | Placebo Part 1, Pexidartinib Part 2 | All Pexidartinib Treated
Number analyzed (Participants) | 61 | 30 | 91
units on a scale
  Baseline: number analyzed (Participants) | 59 | 26 | 85
  Baseline | 5.6 (1.7) | 5.7 (2.3) | 5.6 (1.9)
  Week 25: number analyzed (Participants) | 33 | 18 | 51
  Week 25 | -2.7 (2.2) | -3.0 (3.1) | -2.8 (2.5)
  Week 49: number analyzed (Participants) | 22 | 10 | 32
  Week 49 | -3.5 (1.9) | -2.2 (2.8) | -3.1 (2.3)

16. Other Pre Specified Outcome: Mean Change From Baseline for Worst Pain Numeric Rating Scale Score (NRS) in Participants Receiving Pexidartinib Compared With Those on Placebo by Week 49
Description: The Brief Pain Inventory (BPI) Worst Pain NRS was a 1-item, self-administered questionnaire assessing the "worst" pain in the last 24 hours. The NRS for this item ranged from 0 (no pain) to 10 (pain as bad as you can imagine).
Time Frame: By Week 49
Population: Worst pain was assessed in the ITT population, specifically among the Pexidartinib Part 1, Pexidartinib Part 2; Placebo Part 1, Pexidartinib Part 2; and All Pexidartinib Treated participants. Participants who received Placebo Part 1 only or Pexidartinib Part 2 only were not analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pexidartinib Part 1 and Part 2 | Placebo Part 1, Pexidartinib Part 2 | All Pexidartinib Treated
Number analyzed (Participants) | 61 | 30 | 91
units on a scale
  Baseline: number analyzed (Participants) | 59 | 26 | 85
  Baseline | 5.6 (1.6) | 5.2 (2.5) | 5.5 (1.9)
  Week 25: number analyzed (Participants) | 33 | 18 | 51
  Week 25 | -2.7 (2.2) | -2.6 (3.1) | -2.7 (2.5)
  Week 49: number analyzed (Participants) | 22 | 10 | 32
  Week 49 | -3.3 (1.7) | -2.8 (3.4) | -3.2 (2.3)

17. Other Pre Specified Outcome: Percentage of Participants With Symptomatic, Locally Advanced Tenosynovial Giant Cell Tumor (TGCT) Achieving Complete or Partial Response Based on Tumor Volume Score (TVS) After Receiving Pexidartinib Compared With Those on Placebo by Week 49
Description: Best overall response (CR or PR) was assessed using tumor volume score (TVS) in the ITT population. Tumor Volume Score is a semi-quantitative MRI scoring system that describes tumor mass and is based on 10% increments of the estimated volume of the maximally distended synovial cavity or tendon sheath involved. A tumor that is equal in volume to that of a maximally distended synovial cavity or tendon sheath was scored 10; a score of 0 indicated no evidence of tumor.
Time Frame: By Week 49
Population: Best overall response on Tumor Volume Score was assessed in the ITT population, specifically among the Pexidartinib Part 1, Pexidartinib Part 2; Placebo Part 1, Pexidartinib Part 2; and All Pexidartinib Treated participants. Participants who received Placebo Part 1 only or Pexidartinib Part 2 only were not analyzed..
Measure: Number; unit: Percentage of participants
Arm/Group | Pexidartinib Part 1 and Part 2 | Placebo Part 1, Pexidartinib Part 2 | All Pexidartinib Treated
Number analyzed (Participants) | 61 | 30 | 91
Percentage of participants | 63.9 | 66.7 | 64.8

ADVERSE EVENTS:
Time Frame: Adverse events were monitored throughout the study from the time the participant signed the informed consent form to 28 days after the final treatment dose, up to 71 months.
Groups:
- Pexidartinib (Part 1): Participants received blinded treatment of pexidartinib,1000 mg (5 capsules per day ) for 2 weeks, then 800 mg (4 capsules per day) for 22 weeks
  Pexidartinib: Each capsule contains 200 mg of pexidartinib for oral administration
- Placebo (Part 1): Participants received blinded treatment of matching placebo (5 capsules per day) for 2 weeks, then matching placebo (4 capsules per day) for 22 weeks
  Placebo: Placebo capsule matching pexidartinib capsule for oral administration
- Pexidartinib (Parts 1 and 2): Participants received pexidartinib in Part 1 and in Part 2 at their prescribed dose
  Pexidartinib: Each capsule contains 200 mg of pexidartinib for oral administration
- Placebo (Part 1), Crossover Pexidartinib (Part 2): Participants received placebo in Part 1 and pexidartinib in Part 2 at their prescribed dose
  Pexidartinib: Each capsule contains 200 mg of pexidartinib for oral administration
  Placebo: Placebo capsule matching pexidartinib capsule for oral administration
- All Pexidartinib Treated: All participants who received pexidartinib in Part 1 and Part 2 (placebo crossed over to pexidartinib)
Arm/Group | Pexidartinib (Part 1) | Placebo (Part 1) | Pexidartinib (Parts 1 and 2) | Placebo (Part 1), Crossover Pexidartinib (Part 2) | All Pexidartinib Treated
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/59 | 0/61 | 1/30 | 1/91
Serious Adverse Events (participants affected / at risk) | 8/61 | 1/59 | 12/61 | 9/30 | 21/91
Other Adverse Events (participants affected / at risk) | 60/61 | 55/59 | 61/61 | 30/30 | 91/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pexidartinib (Part 1) (N=61) | Placebo (Part 1) (N=59) | Pexidartinib (Parts 1 and 2) (N=61) | Placebo (Part 1), Crossover Pexidartinib (Part 2) (N=30) | All Pexidartinib Treated (N=91)
Transaminases increased (Investigations) | 1 | 0 | 1 | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0 | 1 | 0 | 1
Hepatic enzyme abnormal (Investigations) | 1 | 0 | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 0 | 1
Adenosquamous carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 1 | 0 | 1
Local swelling (General disorders) | 0 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 1
Hepatoxicity (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Hepatitis A (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Hepatitis E (Infections and infestations) | 1 | 0 | 1 | 0 | 1
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Rectal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pexidartinib (Part 1) (N=61) | Placebo (Part 1) (N=59) | Pexidartinib (Parts 1 and 2) (N=61) | Placebo (Part 1), Crossover Pexidartinib (Part 2) (N=30) | All Pexidartinib Treated (N=91)
Hypertension (Vascular disorders) | 9 (15) | 6 (6) | 14 (24) | 12 (21) | 26 (45)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (7) | 4 (6) | 4 (7) | 2 (2) | 6 (9)
Fatigue (General disorders) | 33 (49) | 21 (26) | 35 (57) | 8 (13) | 43 (70)
Face oedema (General disorders) | 8 (8) | 1 (1) | 9 (11) | 6 (13) | 15 (24)
Oedema peripheral (General disorders) | 8 (9) | 2 (2) | 15 (18) | 9 (11) | 24 (29)
Asthenia (General disorders) | 6 (7) | 3 (5) | 9 (16) | 7 (18) | 16 (34)
Pyrexia (General disorders) | 4 (4) | 1 (1) | 8 (8) | 6 (6) | 14 (14)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 5 (6) | 1 (1) | 6 (7)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 4 (4) | 3 (4) | 7 (8)
Aspartate aminotransferase increased (Investigations) | 24 (48) | 0 (0) | 28 (63) | 6 (11) | 34 (74)
Alanine aminotransferase increased (Investigations) | 17 (44) | 1 (1) | 19 (53) | 7 (13) | 26 (66)
Blood alkaline phosphatase increased (Investigations) | 9 (26) | 0 (0) | 9 (30) | 1 (1) | 10 (31)
Blood lactate dehydrogenase increased (Investigations) | 7 (12) | 0 (0) | 7 (17) | 3 (6) | 10 (23)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 6 (11) | 1 (2) | 7 (13)
Weight increased (Investigations) | 0 (0) | 0 (0) | 3 (4) | 4 (4) | 7 (8)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (2) | 4 (8) | 1 (1) | 5 (9)
Blood creatinine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 6 (16) | 4 (27) | 10 (43)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 1 (2) | 7 (12) | 1 (1) | 8 (13)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 4 (13) | 2 (3) | 6 (16)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 4 (7) | 2 (10) | 6 (17)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (5) | 4 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 4 (6) | 5 (7) | 9 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (4) | 4 (4) | 7 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 4 (4) | 1 (1) | 5 (5)
Dysgeusia (Nervous system disorders) | 15 (24) | 1 (1) | 18 (29) | 7 (10) | 25 (39)
Headache (Nervous system disorders) | 11 (16) | 11 (15) | 15 (25) | 6 (8) | 21 (33)
Dizziness (Nervous system disorders) | 6 (7) | 9 (12) | 10 (14) | 5 (5) | 15 (19)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 6 (7) | 3 (6) | 9 (13)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (7) | 5 (9)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 5 (6)
Periorbital oedema (Eye disorders) | 11 (13) | 1 (1) | 17 (23) | 5 (6) | 22 (29)
Eye oedema (Eye disorders) | 6 (6) | 2 (2) | 6 (6) | 0 (0) | 6 (6)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 3 (5) | 3 (4) | 6 (9)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 5 (5) | 2 (3) | 7 (8)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (6) | 5 (8)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 4 (4) | 4 (4) | 8 (8)
Nausea (Gastrointestinal disorders) | 23 (40) | 24 (27) | 28 (66) | 7 (10) | 35 (76)
Diarrhea (Gastrointestinal disorders) | 13 (17) | 15 (18) | 19 (34) | 10 (23) | 29 (57)
Vomiting (Gastrointestinal disorders) | 12 (16) | 3 (3) | 16 (23) | 3 (3) | 19 (26)
Abdominal pain (Gastrointestinal disorders) | 10 (12) | 6 (8) | 13 (15) | 3 (3) | 16 (18)
Constipation (Gastrointestinal disorders) | 7 (8) | 3 (3) | 10 (13) | 3 (5) | 13 (18)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 2 (2) | 8 (10) | 4 (4) | 12 (14)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 1 (2) | 5 (5) | 3 (5) | 8 (10)
Hair color changes (Skin and subcutaneous tissue disorders) | 41 (46) | 2 (2) | 44 (53) | 25 (39) | 69 (92)
Pruritis (Skin and subcutaneous tissue disorders) | 10 (11) | 2 (2) | 10 (10) | 9 (15) | 19 (25)
Rash (Skin and subcutaneous tissue disorders) | 8 (9) | 3 (4) | 17 (28) | 8 (13) | 25 (41)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (8) | 1 (1) | 10 (17) | 4 (5) | 14 (22)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 6 (10) | 8 (13)
Pruritis generalized (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 6 (7) | 5 (5) | 11 (12)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 5 (6) | 3 (4) | 8 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 6 (6)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (7) | 1 (1) | 6 (8)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (4) | 6 (7)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 3 (4)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (17) | 15 (18) | 19 (29) | 15 (33) | 34 (62)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6) | 3 (3) | 9 (11) | 6 (17) | 15 (28)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 6 (7) | 4 (8) | 10 (15)
Decreased appetite (Metabolism and nutrition disorders) | 10 (13) | 6 (6) | 11 (15) | 3 (4) | 14 (19)
Hypercholesterolemia (Metabolism and nutrition disorders) | 5 (8) | 0 (0) | 7 (20) | 4 (7) | 11 (27)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (6) | 2 (5) | 5 (11)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Nasopharyngitis (Infections and infestations) | 4 (5) | 3 (3) | 5 (7) | 2 (2) | 7 (9)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 8 (11) | 2 (2) | 10 (13)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 5 (9) | 1 (1) | 6 (10)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 4 (4) | 3 (3) | 2 (2) | 5 (5)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 1 (3) | 2 (2) | 3 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 4 (7) | 6 (9)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 4 (6) | 1 (1) | 5 (7)
neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (5) | 5 (6)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (5) | 4 (6)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 2 (2) | 2 (3) | 4 (5) | 6 (8)
Urinary tract infection (Infections and infestations) | 0 (0) | 4 (5) | 2 (2) | 2 (6) | 4 (8)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Lacrimation increased (Eye disorders) | 3 (3) | 0 (0) | 4 (4) | 1 (1) | 5 (5)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 3 (6) | 2 (3) | 5 (9)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 2 (4) | 2 (3) | 4 (7)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 4 (5) | 0 (0) | 4 (5)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 3 (5)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
Enrollment was stopped on 30 Sep 2016; no new participants received the study drug. After Part 1, those who wished to continue were un-blinded; those on placebo were discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT02371369/Prot_SAP_001.pdf